CLINICAL TRIAL: NCT05627830
Title: Ultrasound-Guided Vs Non-Guided Prolotherapy for Internal Derangement of Temporomandibular Joint. a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammad Bader AL-Haj Kheder, Oral & Maxillofacial Surgeon, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111996
Record Dates: First submitted 2022-11-15; First posted 2022-11-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: TMJ Disc Disorder; Ultrasound Therapy; Complications; TMJ; Prolotherapy; Internal Derangement; Clicking Tinnitus; Injection Site; Pain, Chronic; Anterior Disc Displacement; Myofascial Pain Syndrome; Masticatory Muscle
MeSH Terms: conditions — Tinnitus; Chronic Pain; Myofascial Pain Syndromes | interventions — Prolotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Guided Prolotherapy forTreatment of Internal Derangement of TMJD. (Experimental): Injection procedure in TMJ Space guided by ultrasound probe the injection materials will be composition of ( !0% Dextrose ) + (Saline ) + (2% Lidocaine, plain anesthesia ).
  The intervention procedure will done after TMJ MRI assessment for patients who have anterior disc displacement with reduction (DDWR)
  Interventions: Procedure: Prolotherapy
- Non-Guided Ultrasound ( Blind) Prolotherapy for Treatment of Internal Derangement of TMJD. (Active Comparator): Injection procedure in TMJ Space by anatomical land mark (blindly), and we also call it ( conventional prolotherapy ) the injection materials will be composition of ( !0% Dextrose ) + (Saline ) + (2% Lidocaine, plain anesthesia ).
  The intervention procedure will done after TMJ MRI assessment for patients who have anterior disc displacement with reduction (DDWR)
  Interventions: Procedure: Prolotherapy

INTERVENTIONS:
Procedure: Prolotherapy — Prolotherapy is an injection treatment used to relieve pain. And for Cellular Regeneration

SUMMARY:
Ultrasound Guided Versus Non-Guided Prolotherapy for Treatment of Internal Derangement of Temporomandibular joint.

Rationale for conducting the research:

The most critical cause for guided prolotherapy is to specify the accurate location of glenoid fossa and the disc space while prolotherapy procedure, and to adjust the needle insertion to according to articular eminence, mandibular condyle, and intra-articular space as anatomical variations. The vibration of ultrasound waves generates a heat so there is a thermal effective for prolotherapy effusion in the TMJ space.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with TMD - internal derangement with symptomatic clicking pain, according to RDC (Research diagnostic criteria for TMJD) sheet .
2. Muscles spasm causing TMDs.
3. Patients who failed to improve on conservative measures or highly hyperactivity patients.
4. Female and male patients age range from 20 to 60 years old.

Exclusion Criteria:

1. Patients who refused to be included in the research.
2. Patients with a systemically diseases or inflammation whether local or generalized.
3. Patients with bleeding disorders.
4. Patients with unknown dextrose allergy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | Change from Baseline VAS at 4 weeks ( lower score means better outcome)
  psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients
visual analogue scale | VAS change at 2 months ( lower score means better outcome )
  psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients

CONTACTS AND LOCATIONS:
Locations (1):
- CairoU, Cairo, Al Manial, Old Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The data of volunteers will be shared with the doctors supervising the thesis research to assess the status and results of the scientific research